CLINICAL TRIAL: NCT01446341
Title: A Pilot Study Towards a Randomized Clinical Trial of Cast Immobilization Versus Functional Therapy for Acute, Severe Lateral Ankle Sprains
Brief Title: Cast Immobilization Versus Functional Therapy for Acute, Severe Lateral Ankle Sprains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Workers' Compensation Board of BC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H11-01150
Record Dates: First submitted 2011-08-19; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Ankle Sprain
Keywords: Ankle sprain; Functional rehabilitation; Immobilization
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immobilization (Active Comparator): 50 patients will be randomly assigned to have their lateral ankle sprain immobilized in a below knee cast
  Interventions: Procedure: Below knee plaster casting
- Functional Rehabilitation (Active Comparator): 50 patients will be randomly assigned to a functional rehabilitation program for their lateral ankle sprain
  Interventions: Procedure: Functional rehabilitation

INTERVENTIONS:
Procedure: Below knee plaster casting — Subjects will be randomly assigned to either immobilization of their lateral ankle sprain with a below knee cast or to enter a functional rehabilitation program
  Arms: Immobilization
Procedure: Functional rehabilitation — Subjects will be randomly assigned to either immobilization of their lateral ankle sprain with a below knee cast or to enter a functional rehabilitation program
  Arms: Functional Rehabilitation

SUMMARY:
Acute, severe lateral ankle sprains are estimated to comprise between 3-5% of emergency department visits and are the most common musculoskeletal injury in the physically active population. Although the current accepted treatment of ankle sprains is to encourage early mobilization with functional rehabilitation, there is little high-quality evidence directing this clinical practice.

This pilot study is to:

* provide quantitative data for estimation of mean outcome scores and standard deviations to allow subsequent sample size calculations
* evaluate the feasibility of the proposed study design
* assess patient enrollment issues specific to randomization into an active rehabilitation program compared to below knee immobilization.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* meet clinical criteria for unilateral grade II-III ankle sprains (inability to weight bear)

Exclusion Criteria:

* bony injury on x-ray or computed tomography
* contraindications to recurrent icing
* high risk of deep-vein thrombosis
* injury greater than 3 days old
* ongoing recovery from previous acute ankle sprain
* age greater than 60
* non-English speaking patients, those patients unable to provide informed consent or patients with insufficient contact information for follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Foot and Ankle Outcome Score (FAOS)measured at 1 and 3 months. | Measured at 0, 1, and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Rose, MD, PhD, Principal Investigator — University of British Columbia - Vancouver Coastal Health Research Institute